CLINICAL TRIAL: NCT02328534
Title: Novel Approach of Semen Preparation to Improve ICSI Outcome.
Brief Title: Semen Processing for ICSI Using Swim-down and Density Gradient Methods
Status: Completed | Type: Observational
Sponsor: Ahmad Mustafa Mohamed Metwalley (Other)
Responsible Party: Sponsor-Investigator, Ahmad Mustafa Mohamed Metwalley, Novel Approach of Semen Preparation to Improve ICSI Outcome, Al Baraka Fertility Hospital
Organization: Al Baraka Fertility Hospital (Other)
Other Study IDs: AlBarakaSD1
Record Dates: First submitted 2014-12-28; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Infertility
Keywords: ICSI/IVF; Semen processing; Semen preparation; Swim down; Density gradient; Silica solution
MeSH Terms: conditions — Infertility | interventions — Pregnancy Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Semen samples Embryos processed after ICSI and IVF cycles.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Density Gradient semen: ICSI Cases processed using DG semen processing and evaluated by
  Blastocyst Formation Rate Blastocyst Rate Pregnancy Rate
  Interventions: Behavioral: Blastocyst Formation Rate; Procedure: Blastocyst Rate; Procedure: Pregnancy Rate
- Swimming down semen: ICSI Cases processed using SD semen processing and evaluated by
  Blastocyst Formation Rate Blastocyst Rate Pregnancy Rate
  Interventions: Behavioral: Blastocyst Formation Rate; Procedure: Blastocyst Rate; Procedure: Pregnancy Rate

INTERVENTIONS:
Behavioral: Blastocyst Formation Rate — Embryos developed at Day3 cultures, are continued for Day5 culture tho reach blastocyst stage. The percentage of blastocyst produced from cleaved embryos to be evaluated ar rate.
  The evaluation with doe one time using Density Gradient semen one time and Swimming down semen another time.
  Other Names: Blastocyst developed form cleaved embryos
Procedure: Blastocyst Rate — Day 5 embryo transfer achieved pregnancy are compared with total embryo transfer cases at Day5.
  The evaluation with doe one time using Density Gradient semen one time and Swimming down semen another time.
  Pregnancy confirmed with day 12 after Et and repeated with 48 hours after 1st exam.
  Other Names: Pregnancey produced formblastocyst embryo transfer
Procedure: Pregnancy Rate — All pregnancy achieved from all ET. Pregnancy confirmed with day 12 after Et and repeated with 48 hours after 1st exam.
  The evaluation with doe one time using Density Gradient semen one time and Swimming down semen another time.
  Other Names: Pregnancy achieved after all ET

SUMMARY:
The investigators evaluate the feedback of using swim down semen processing method during preparation for ICSI and compare the results of pregnancy and embryos quality with the cases used density gradient method for their semen processing.

DETAILED DESCRIPTION:
There is different semen processing method, in this study we compared the ICSI output when the investigators used one method with higher separation method and minimum sperm stress or physical interface as swimming down using 100 % silica solution, with other more stressful procedure with high selection power as density gradient.

The routine used method as density gradient (DG) includes about 30 min centrifugation at 1200 RPM, and more working steps with more handling procedures. According to many references the investigators can approve that it is method to be indicated with all cases particularly with those severely decreases semen number or motility.

Using 100 % silica solution for semen processing used for ICSi, shews lesser centrifugation time and minimum processing procedures. As swimming down time is about 30 min followed by 5 min washing and finalized with other 3 minutes last wash. For that total interfering physical action is about 8 minutes compared with 30 min with DG method.

In swimming down we are using the natural sperm behavior and own swimming power for separate itself from other seminal components. As well as only the one normally structure and motility direction the only can penetrate the interface surface of silica solution and swim inside higher density matrix using its speed and power.

ELIGIBILITY:
Inclusion Criteria: all semen samples fresh or frozen that has,

* Cases have semen examination criteria fall within WHO 2010 standards of count
* Cases have semen examination criteria fall within WHO 2010 standards of motility
* Cases have semen examination criteria with all types of abnormal forms
* Cases produced more than 4 mature oocytes (M2) and more

Exclusion Criteria:

* Cases have semen examination criteria with motility less than 5%
* Cases have semen examination criteria with count less than 1.0 million
* Cases with TESE, TESA and EPSA, both fresh and frozen
* Cases produced less than 4 mature oocytes (M2)

Ages: 20 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Cases collected were submitted for ART treatment using ICSI/IVF procedures. In two different IVF clinics at Manama-Bahrain and Sohag-Egypt. The groups of about 890 couple prepared for treatment.
Sampling Method: Probability Sample
Enrollment: 890 (Actual)
Dates: Start 2007-03; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Total Pregnancy Rate | 3 Years
  Percentage of Pregnancies developed after embryo transfer, for maternal age less than 38 years old.

SECONDARY OUTCOMES:
Blastulation Rate (BR) | 3 years
  Percentage of blastocyst embryos produced from cleaved embryos, for maternal age less than 38 YO.
Blastocyst formation Rate (BFR) | 3 Years
  Developed embryos developed to Blastocyst stage from cleaved embryos.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M Metwalley, Ms. Genetics, Study Director — Adliyah
Locations (2):
- Al Baraka Fertility Hospital, Manama, Adliyah, Bahrain
- Ibn Sina IVF Center- Ibn Sina Hospital, Sohag, Sohag Governorate, Egypt

REFERENCES:
- [Result] Malvezzi H, Sharma R, Agarwal A, Abuzenadah AM, Abu-Elmagd M. Sperm quality after density gradient centrifugation with three commercially available media: a controlled trial. Reprod Biol Endocrinol. 2014 Dec 2;12:121. doi: 10.1186/1477-7827-12-121. PMID 25466430
- See also: Density Gradient procedures description — http://www.springerprotocols.com/Abstract/doi/10.1007/978-1-62703-038-0_19